CLINICAL TRIAL: NCT04870788
Title: Cultural Adaptation of a Mindfulness-Based Intervention for Latino Cancer Patients and Their Caregivers
Brief Title: Mindfulness-Based Intervention for Latino Cancer Patients and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1070; NCI-2021-02774 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1070 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-12; First posted 2021-05-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Neoplasm
MeSH Terms: interventions — Mindfulness; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (mindfulness program) (Experimental): Patients and their partners participate together in mindfulness program over 60 minutes consisting of meeting with a mindfulness coach to build awareness of thoughts, emotions, feelings, and sensations QW for 4 weeks.
  Interventions: Behavioral: Mindfulness Relaxation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Group II (mindfulness waitlist)
- Group II (mindfulness program) (Experimental): Patients and their partners participate separately in mindfulness program over 60 minutes consisting of meeting with a mindfulness coach to build awareness of thoughts, emotions, feelings, and sensations QW for 4 weeks.
  Interventions: Behavioral: Mindfulness Relaxation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Group II (mindfulness waitlist)

INTERVENTIONS:
Behavioral: Mindfulness Relaxation — Participate in mindfulness program
  Other Names: MBSR; Mindful Meditation; Mindfulness Meditation; Mindfulness-Based Stress Reduction
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Group II (mindfulness waitlist) — Patients and their partners participate in mindfulness program together or separately, depending on their preference, as in Group I beginning 12 weeks after starting the study and completing the third study visit.

SUMMARY:
This clinical trial develops effective and appropriate mindfulness-based interventions that help meet the needs of Latino cancer patients and their family caregivers. Mindfulness-based interventions focus on building awareness of thoughts, emotions/feelings, and the sensations. This study may help improve mental well-being and reduce stress and anxiety associated with having cancer or with a family member's cancer diagnosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Systematically and culturally adapt a mindfulness-based intervention to improve psychological wellbeing in Latino patients with advanced cancer and their family caregivers.

II. Evaluate the feasibility of the adapted mindfulness-based intervention and overall study procedures in Latino patient-family caregiver dyads.

SECONDARY OBJECTIVE:

I. Determine the effects of the adapted mindfulness-based intervention on the secondary outcomes of patient and caregiver psychological distress, quality of life (QOL), and patient cancer symptoms, compared to a waitlist control.

OUTLINE: Patients and their partners are randomized to 1 of 32 groups.

GROUP I: Patients and their partners participate in mindfulness program together over 60 minutes consisting of meeting with a mindfulness coach to build awareness of thoughts, emotions, feelings, and sensations 1 time per week (QW) for 4 weeks.

GROUP II: Patients and their partners participate in mindfulness program separately over 60 minutes consisting of meeting with a mindfulness coach to build awareness of thoughts, emotions, feelings, and sensations 1 time per week (QW) for 4 weeks.

GROUP III: Patients and their partners participate in mindfulness program either separately or together, depending on participants' preferences, as in Group I beginning 12 weeks after starting the study and completing the third study visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a stage III-IV solid tumor
* On active treatment
* Self-identify as Hispanic/Latino
* ECOG (Eastern Cooperative Oncology Group) performance status of =< 2
* Willing to participate in the study with a family caregiver (e.g., spouse, adult child) with whom they currently reside and who consents to participate

Exclusion Criteria:

* At least 18 years old
* Able to speak English or Spanish
* Have access to the internet
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall accrual | Up to 12 weeks
  Will calculate means, frequencies, and 90% confidence intervals (CIs), as applicable.
Attrition | Up to 12 weeks
  Will calculate means, frequencies, and 90% CIs, as applicable.
Adherence | Up to 12 weeks
  Will calculate means, frequencies, and 90% CIs, as applicable.
Acceptability | Up to 12 weeks
  Will calculate means, frequencies, and 90% CIs, as applicable.

SECONDARY OUTCOMES:
Patient and caregiver psychological distress | At 6 and 12 weeks
  Will examine means, standard deviations (SDs), and distributions of survey measures for ceiling/floor effects and restrictions in range and examine change over time.
Quality of life questionnaire | At 6 and 12 weeks
  Will examine means, SDs, and distributions of survey measures for ceiling/floor effects and restrictions in range and examine change over time.
Patient cancer symptoms | At 6 and 12 weeks
  Will examine means, SDs, and distributions of survey measures for ceiling/floor effects and restrictions in range and examine change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin Strong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org